CLINICAL TRIAL: NCT00817284
Title: A Randomized Phase II Trial With Bevacizumab, Irinotecan and Cerebral Radiotherapy Versus Bevacizumab, Temozolomide and Cerebral Radiotherapy as First Line Treatment for Patients With Glioblastoma Multiforme
Brief Title: Bevacizumab and Irinotecan or Bevacizumab and Temozolomide With Concomitant Radiotherapy for Primary Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ulrik Lassen (Other)
Responsible Party: Sponsor-Investigator, Ulrik Lassen, MD., PH.D. Chief Physician, Phase I Unit, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIBT-01
Record Dates: First submitted 2008-12-08; First posted 2009-01-06 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Glioblastoma Multiforme
Keywords: Newly diagnosed patients with glioblastoma multiforme.; Performance status 0-2.
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Irinotecan; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm I (Experimental): Bevacizumab + Irinotecan and concomitant radiotherapy
  Interventions: Drug: bevacizumab and Irinotecan and radiotherapy
- Arm II (Experimental): Bevacizumab and Temozolomide and concomitant radiotherapy
  Interventions: Drug: Bevacizumab and Temozolomide and radiotherapy

INTERVENTIONS:
Drug: bevacizumab and Irinotecan and radiotherapy — * Bevacizumab 10 mg/kg is administered on days 1 and 15.
  * Irinotecan:
  * Irinotecan 125 mg/m2 is administered on days 1 and 15 to patients NOT receiving enzyme-inducing antiepileptic drugs (EIAED).
  * Irinotecan 340 mg/m2 is administered on days 1 and 15 to patients receiving EIAEDs.
  * During concomitant chemoradiotherapy, bevacizumab and irinotecan are given in the same doses and schedules as before and after chemoradiotherapy.
  Radiotherapy is delivered during 3rd and 4th cycle of chemotherapy and consists of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily five days per week (Monday to Friday) over a period of six weeks for a total dose of 60 Gy.
  Arms: arm I
Drug: Bevacizumab and Temozolomide and radiotherapy — Bevacizumab 10 mg/kg is administered on days 1 and 15. Temozolomide dosing before start concomitant chemoradiotherapy: 150 mg/m2/day on days 1-5 during the first 28 days treatment cycle, then 200 mg/m2/day on the subsequent cycles until radiotherapy.
  Temozolomide administered concomitantly with the radiotherapy: Temozolomide 75 mg/m2/day for 7 days per week is administered on each day of radiotherapy.
  After completed chemoradiotherapy, temozolomide is dosed and administered as it was prior to start chemoradiotherapy, i.e. temozolomide 200 mg/m2/day on days 1-5 out of a 28 days schedule, taking into consideration any previous dose-reductions already made.
  Radiotherapy is delivered during 3rd and 4th cycle of chemotherapy and consists of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily five days per week (Monday to Friday) over a period of six weeks for a total dose of 60 Gy.
  Arms: Arm II

SUMMARY:
Significant activity (radiographic response rates of approximately 60%) has recently been demonstrated in phase II studies in patients with relapsed GBM from the combined use of Irinotecan (CPT-11) and bevacizumab. The 6-month progression-free survival rate is 30% and median survival duration is 9 months. The current first line therapy of GBM patients following initial surgical resection/debulking is the concomitant use of cerebral radiotherapy and the orally available alkylating agent temozolomide, followed by temozolomide for 6 months post-radiotherapy.

Considering the significant activity of the combination of Bevacizumab + irinotecan in patients with recurrent GBM, and considering the activity of temozolomide in GBM, it is proposed that the combination of Bevacizumab + Temozolomide may also be an active regimen. Bevacizumab + Temozolomide display non-overlapping toxicity clinically and thus their combined use without significant dose-reductions seems rational.

The toxicity from the combined use of the two drugs prior to radiotherapy, as well as the toxicity when administered together with radiotherapy, is evaluated.

This study will try to identity whether Bevacizumab and Irinitecan or Bevacizumab and Temozolomide should be the experimental arm in future phase III comparison with standard care with concomitant Temozolomide and radiotherapy.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Histological verified primary glioblastoma multiforme
* No prior therapy for GBM, except for primary surgical resection or biopsy
* PS 0-2
* Age > 18
* Expected survival > 3 months
* Adequate liver, renal and bone-marrow function, determined as:

  * Thrombocytes > 100 x 109/liter
  * Hemoglobin >6.2 mmol/liter
  * Leukocytes > 3 x 109/liter
  * Neutrophil granulocytes > 1.5 x 109/liter
  * ASAT and/or ALAT < 3 x upper normal limit
  * Bilirubin < 1.5 x upper normal limit
  * Serum-creatinin < upper normal limit or glomerular filtration rate >60 ml/min (corrected for age) determined by measurement of clearance of Cr-EDTA
  * APTT < upper normal limit
  * INR < upper normal limit
* Fertile women of childbearing age must use proper anti-conception (oral contraceptives, IUD and/or condom). Fertile men must use condom
* No sign of cerebral bleeding on cerebral MR-scanning at baseline.

Exclusion criteria:

* Previous therapy of GBM, including radiotherapy and the use of biological " targeted" drug, e.g. drugs targeted against the VEGF- or EGFR pathway
* Concurrent use of medication that can affect the interpretation of the results from the study, e.g. use of immunosuppressive drugs, except corticosteroids
* Conditions (medical, social or physical) that may compromise proper information and/or follow-up
* Other concurrent or previous cancer within 5 years, except adequately treated basal or planocellular skin cancer, or cervical carcinoma in situ
* Significant heart disease (according to the New York Heart Association class II or more severe), clinically significant arrhythmia or unstable angina pectoris/acute myocardial infarction within last 6 months
* Clinical significant peripheral arterial disease
* Known or suspected disorders of coagulation or concurrent therapy with ASA, NSAID or clopidogrel
* Major surgery, open biopsy or greater trauma, or expectations thereof, within 28 days prior to start of therapy
* Minor surgery or needle biopsy, or expectations thereof, within 7 days prior to start of therapy
* Known or suspected abdominal fistulas, gastrointestinal perforations or intra-abdominal abscesses within 6 months prior to start of therapy
* Chronic inflammatory intestinal disease and/or intestinal obstruction
* Known or active HIV or Hepatitis B/C infection
* Concurrent ongoing significant infection or diabetes mellitus not adequately controlled medically
* Clinically significant non-healing ulcers
* Active ventricular or duodenal ulcers within 6 months prior to start of therapy
* Recent bone-fracture (<3 months)
* Pregnancy or lactation
* Need for systemic anticoagulant therapy at time of start of therapy
* Blood pressure > 150/100 mmHg (patients are allowed to receive proper antihypertensive medication)
* Proteinuria ≥ 1 gram/day
* Known allergy toward irinotecan (or related substance) or vehicle
* Known allergy toward temozolomide (or related substance) or vehicle
* Known allergy toward bevacizumab (or related substance) or vehicle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate according to McDonald criteria | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Århus Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense Hospital, Odense